CLINICAL TRIAL: NCT03506750
Title: Different Day Regimes of Preoperative CONbercept Administration on CytokinEs of Proliferative Diabetic Retinopathy Patients Undergoing Vitrectomy: a Prospective Randomized Controlled Clinical Trial (CONCEPT)
Brief Title: Day Regimes of CONbercept on CytokinEs of PDR Patients Undergoing Vitrectomy - Trial (CONCEPT)
Acronym: CONCEPT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zizhong Hu, Dr., The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CONCEPT
Record Dates: First submitted 2018-03-09; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Proliferative Diabetic Retinopathy; VEGF Overexpression
Keywords: Conbercept; PLGF
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- IVC-1day (Experimental): patients with proliferative diabetic retinopathy receiving IVC 1 days before surgery
  Interventions: Drug: IVC; Procedure: Blood and aqueous humor at the time of IVC; Procedure: Collect blood, aqueous humor, and initial vitreous at the time of surgery.
- IVC-2day (Experimental): patients with proliferative diabetic retinopathy receiving IVC 2 days before surgery
  Interventions: Drug: IVC; Procedure: Blood and aqueous humor at the time of IVC; Procedure: Collect blood, aqueous humor, and initial vitreous at the time of surgery.
- IVC-3day (Experimental): patients with proliferative diabetic retinopathy receiving IVC 3 days before surgery
  Interventions: Drug: IVC; Procedure: Blood and aqueous humor at the time of IVC; Procedure: Collect blood, aqueous humor, and initial vitreous at the time of surgery.
- IVC-4day (Experimental): patients with proliferative diabetic retinopathy receiving IVC 4 days before surgery
  Interventions: Drug: IVC; Procedure: Blood and aqueous humor at the time of IVC; Procedure: Collect blood, aqueous humor, and initial vitreous at the time of surgery.
- IVC-5day (Experimental): patients with proliferative diabetic retinopathy receiving IVC 5 days before surgery
  Interventions: Drug: IVC; Procedure: Blood and aqueous humor at the time of IVC; Procedure: Collect blood, aqueous humor, and initial vitreous at the time of surgery.
- IVC-6day (Experimental): patients with proliferative diabetic retinopathy receiving IVC 6 days before surgery
  Interventions: Drug: IVC; Procedure: Blood and aqueous humor at the time of IVC; Procedure: Collect blood, aqueous humor, and initial vitreous at the time of surgery.
- IVC-7day (Experimental): patients with proliferative diabetic retinopathy receiving IVC 7 days before surgery
  Interventions: Drug: IVC; Procedure: Blood and aqueous humor at the time of IVC; Procedure: Collect blood, aqueous humor, and initial vitreous at the time of surgery.
- IVC-sham (Sham Comparator): patients with proliferative diabetic retinopathy receiving sham IVC
  Interventions: Procedure: Collect blood, aqueous humor, and initial vitreous at the time of surgery.; Procedure: IVC-sham
- non-DR (Placebo Comparator): patients with other retinopathy (idiopathic macular hole or epiretinal membrane)
  Interventions: Procedure: Collect blood, aqueous humor, and initial vitreous at the time of surgery.

INTERVENTIONS:
Drug: IVC — Patients with PDR will receive intravitreal injection of conbercept (0.5 mg/0.05 mL; Chengdu Kanghong Biotech, Inc., Chengdu, Sichuan, China) in the inferior-temporal sector 4 mm from the sclerocorneal limbus before pars plana vitrectomy (PPV) surgery.
  Arms: IVC-1day; IVC-2day; IVC-3day; IVC-4day; IVC-5day; IVC-6day; IVC-7day
Procedure: Blood and aqueous humor at the time of IVC — Initial blood and aqueous humor will be harvested at the time of IVC.
  Arms: IVC-1day; IVC-2day; IVC-3day; IVC-4day; IVC-5day; IVC-6day; IVC-7day
Procedure: Collect blood, aqueous humor, and initial vitreous at the time of surgery. — Blood, aqueous humor, and vitreous will be collected at the time of surgery.
Procedure: IVC-sham — Patients with PDR will receive sham intravitreal injection of conbercept in the inferior-temporal sector 4 mm from the sclerocorneal limbus 4 days before PPV surgery.
  Arms: IVC-sham

SUMMARY:
Patients with proliferative diabetic retinopathy requiring surgical intervention will receive a pre-operative injection of Conbercept. Patients will be recruited into different groups according to variable time intervals (1 to 7 days) between intravitreous injection and surgery. At initial, pre-injection aqueous humor and blood sample will be collected in order to provide baseline VEGF-A, -B, placental growth factor (PIGF), and other cytokine levels. At the onset of the vitrectomy, a second aqueous humor, blood, and vitreous sample will be taken to obtain intra-operative levels of , VEGF-A, -B, PIGF, and other cytokine levels.

DETAILED DESCRIPTION:
Proliferative diabetic retinopathy (PDR), characterized by neovascularization and ﬁbrous proliferation, is a severe and common complication of diabetes mellitus (DM). Persistent vitreous hemorrhage (VH) caused by neovascularization and tractional retinal detachment (TRD) caused by ﬁbrous proliferation can lead to permanent vision loss or even blindness, which are the most common indications for surgical intervention.

As neovascularization is the basal pathophysiological change of PDR and vascular endothelial growth factor (VEGF) has been acknowledged as primary angiogenesis factor, the preoperative adjunctive use of VEGF blockade is rationally proposed. The anti-VEGF drugs have been reported to be effective in bringing about regression of retinal neovascularization, shortening surgical duration, avoiding risk of iatrogenic retinal hole and secondary operation for the recurrent VH.

Conbercept (KH902) is a newly developed anti-VEGF drug and has been applied in clinic. Because of its additional binding domain of VEGFR-2, conbercept can bind to all isoforms of VEGF-A, VEGF-B, and placental growth factor (PLGF). A number of studies have presented its high affinity in the treatment of fundus diseases such as wet age-related macular degeneration (wet-AMD), macular edema secondary to retinal vein occlusion[8] and diabetic retinopathy. Also, recent randomized controlled trials have shown its protective effect of conbercept for the surgical treatment of PDR.

Although the overwhelming clinical evidence supports the anti-VEGF drugs as the preoperative adjuncts for PDR, the optimal duration between anti-VEGF injection and surgical intervention has not yet reached a consensus. Longer duration is related to higher incidence of the development or progression of TRD. It might provide clues by investigation of the pattern of cytokine changes in humor aqueous, vitreous, and blood. No studies have been done to date in patients with PDR to quantify the reduction of intravitreal VEGF-A, -B, PLGF or other cytokines levels in these patients following intravitreal Conbercept injection or to evaluate the effects of VEGF or PIGF blockade on the neovascular regression and surgical outcome in patients with extensive diabetic proliferative neovascularization.

The goal of this study is to quantify the reduction of changes of VEGF-A, -B, PLGF levels in patients receiving r pre-operative intravitreal Conbercept after variable time intervals (1, 2, 3, 4, 5, 6, 7 days).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Type 1 or 2 diabetes
* PDR patients requiring surgical intervention for complications of vitreous hemorrhage or traction retinal detachment and pre-operative IVC treatment.
* women postmenopausal for 12 months before the study, surgically sterile, or not pregnant and on effective contraception.

Exclusion Criteria:

* previous retinal vein occlusion.
* any intraocular surgery within the previous 12 months.
* myopia of > or = to 8 diopters.
* active ocular or periocular infection
* treatment with an investigational agent for any condition 60 days prior to enrollment.
* evidence of severe cardiac disease.
* clinically significant peripheral vascular disease (previous surgery, amputation, or symptoms of claudication)
* uncontrolled hypertension (treated systolic blood pressure > 155 mmHg or diastolic blood pressure > 95 mmHg)
* stroke within the preceding 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-06-03 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of intraocular VEGF and PLGF of patients with proliferative diabetic retinopathy post-IVC (intravitreous injection of Conbercept). | 1-7 days

SECONDARY OUTCOMES:
Changes of serum angiogenesis-related pro-cytokines in patients with proliferative diabetic retinopathy | 1-7 days
Changes of intraocular and serum proﬁbrotic cytokines in patients with proliferative diabetic retinopathy post-IVC. | 1-7 days
Changes of intraocular and serum inflammatory cytokines in patients with proliferative diabetic retinopathy post-IVC. | 1-7 days
Vitreous concentration of Conbercept | 1-7 days
  Detection of Vitreous concentration of the drug of Conbercept (Conbercept is a kind of fusion protein)
Effect of IVC on surgery time of surgery | Surgery day
  surgery time of vitrectomy
Effect of IVC on intraoperative complication of surgery | Surgery day
  Record the intraoperative complication: bleeding and iatrogenic retinal hole when surgically removing the proliferative membranes.
Effect of IVC on regression of neovascularization on vitreous fibrovascular membrane with optic coherence tomography angiography (OCTA) | 1 to 7 days
  OCTA monitor the changes of neovascularization on vitreous fibrovascular membrane after IVC and before surgery
Effect of IVC on postoperative visual acuity | 1 to12 months
  Best-corrected visual acuity postoperatively
Effect of IVC on postoperative complications | 1 to12 months
  Record number of patient with vitreous re-bleeding and iris neovascularization postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Qinghuai Liu, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Chen DY, Sun NH, Chen X, Gong JJ, Yuan ST, Hu ZZ, Lu NN, Korbelin J, Fukunaga K, Liu QH, Lu YM, Han F. Endothelium-derived semaphorin 3G attenuates ischemic retinopathy by coordinating beta-catenin-dependent vascular remodeling. J Clin Invest. 2021 Feb 15;131(4):e135296. doi: 10.1172/JCI135296. PMID 33586674